CLINICAL TRIAL: NCT06119035
Title: Insulin Modelling Based on Plasma Glucose Measures Via a Minimally-Invasive Glucose Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Chun Yip James Chan, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-100
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Water

STUDY DESIGN:
Intervention Model Description: The study will be carried out as a single-arm, unblinded, intervention study. The total duration of the study is 4 hours and 30 minutes over one day, excluding screening and enrolment time (up to 1 hour).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prediabetic (Other): n=10, single dose of 75 grams glucose in 200ml water
  Interventions: Other: Single dose of 75 grams glucose in 200ml water

INTERVENTIONS:
Other: Single dose of 75 grams glucose in 200ml water — Consume single dose of 75 grams glucose in 200ml water

SUMMARY:
The study aims to evaluate insulin as a potential biomarker for prediabetes in Singapore Chinese subjects.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2DM) in Singapore is expected to increase from 400,000 to 1,000,000 individuals by 2050, resulting in nearly US$2 billion in economic costs. Pre-diabetes is defined as an intermediate state of hyperglycemia where blood glucose levels are elevated but are below the diagnostic levels of diabetes. In Singapore, approximately 1 in 7, or 430,000 residents are estimated to be pre-diabetic, and globally this number is estimated at 7.3% of adults (equivalent to 352.1 million individuals). Up to 70% of pre-diabetics eventually develop overt T2DM; however, pre-diabetes may be reversible with early detection, providing a window for opportune disease interception.

While blood glucose is currently used to detect pre-diabetes, homeostatic mechanisms can maintain normal blood glucose levels and mask the detection of pre-diabetes until overt hyperglycemia is exhibited. In contrast, numerous studies have demonstrated that insulin levels increase markedly in pre-diabetes, even as marginal changes are observed in glucose levels. In this study, the investigator aims to determine if dynamic insulin levels observed during an oral glucose tolerance test are more sensitive than glucose alone in detecting prediabetes in a Singapore Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-60
* Chinese ethnicity
* Male or female
* Adequate fluency in the English language to understand the informed consent process, study instructions and study assessments.
* Sufficient vision and hearing to complete the study procedures
* Willing and able to participate and to give written informed consent

Exclusion Criteria:

* Diabetes diagnosis based on HbA1c ≥ 6.5%, and fasting plasma glucose ≥ 7.0 mmol/L
* Past (<3 months prior to the study) or current major metabolic, endocrine, gastrointestinal or cardiovascular disease
* Individuals diagnosed with non-alcoholic fatty liver disease
* Women diagnosed with polycystic ovary syndrome
* Major surgery in the past 2 months
* Past (<1 month prior to the study) or current use of prescription, over the counter or traditional medication that may influence metabolic or gastrointestinal functioning
* Presence or past history of alcohol or drug addiction
* Smoking
* Pregnant or lactating
* Alcohol intake >1 units per day
* Body Mass Index <18.5 kg/m2 or ≥30 kg/m2
* Member of the research team or their immediate family members

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Glycated Haemoglobin (HbA1c) levels will be analyzed | 0 minutes
  Blood samples will be collected at 1 time point before intervention administration
Insulin levels will be analyzed | 4 hours 30 minutes
  Blood samples will be collected at 17 time points
Glucose levels will be analyzed | 4 hours 30 minutes
  Blood samples will be collected at 17 time points

SECONDARY OUTCOMES:
Serum samples | up to 3 years
  Serum samples will be frozen for additional future analysis

CONTACTS AND LOCATIONS:
Overall Officials: James Chan, PhD, Principal Investigator — Singapore Institute of Food and Biotechnology Innovation (SIFBI), A*STAR
Locations (1):
- Human Development Research Centre, SICS, A*STAR, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ow Yong LM, Koe LWP. War on Diabetes in Singapore: a policy analysis. Health Res Policy Syst. 2021 Feb 8;19(1):15. doi: 10.1186/s12961-021-00678-1. PMID 33557840
- [Background] Wang Q, Jokelainen J, Auvinen J, Puukka K, Keinanen-Kiukaanniemi S, Jarvelin MR, Kettunen J, Makinen VP, Ala-Korpela M. Insulin resistance and systemic metabolic changes in oral glucose tolerance test in 5340 individuals: an interventional study. BMC Med. 2019 Nov 29;17(1):217. doi: 10.1186/s12916-019-1440-4. PMID 31779625
- [Result] Tan KW, Dickens BSL, Cook AR. Projected burden of type 2 diabetes mellitus-related complications in Singapore until 2050: a Bayesian evidence synthesis. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e000928. doi: 10.1136/bmjdrc-2019-000928. PMID 32184203
- See also: Describes Singapore's War on Diabetes, the Ministry of Health (MOH) is studying measures to better support pre-diabetic persons in managing their condition. — http://www.moh.gov.sg/news-highlights/details/ministry-of-health-studying-measures-to-better-support-persons-with-pre-diabetes